CLINICAL TRIAL: NCT04448743
Title: Role of Circulating Microparticles in Covid-19 Infection
Brief Title: Role of Microparticles in Covid-19 Infection
Acronym: MICO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7829
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: microparticles; microvesicles; vessel; vasculature; endothelium; coagulation; thrombosis
MeSH Terms: conditions — COVID-19; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Covid-19 patients
  Interventions: Other: Blood sample
- patients with coronary artery disease
  Interventions: Other: Blood sample
- healthy volunteers
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 20 Ml blood sample

SUMMARY:
Among the distinctive features of Covid-19, numerous reports have stressed the importance of vascular damages associated with coagulopathy onset. Microparticles (MPs) shed by apoptotic/stimulated cells are reliable markers of vascular damage released upon pro-inflammatory conditions and behave as active participants in the early steps of clot formation. In addition, MPs carry ACE1 and ACE2, the cell-entry receptor for SARS-Cov2 in the vasculature and up-regulate ACE1 expression in neighbouring endothelial cells. This may contribute to unopposed angiotensin II accumulation which further exacerbate tissue injury and promote both inflammation and thrombosis. The aim of the study is to evaluate the impact of circulating MPs on ACE2 expression, the cell-entry receptor for SARS-Cov2 on endothelial cells.

DETAILED DESCRIPTION:
Circulating MPs will be isolated from Covid-19 patients with lupus anticoagulant, from coronary artery diseases patients and from healthy volunteers without cardiovascular risk factors. Quantification of MPs will be realized by prothrombinase assay. Primary endothelial cells (ECs) from porcine coronary artery or porcine pulmonary artery will be isolated and cultured. ECs will be exposed to circulating MPs. Phenotypical changes (ACE2 expression, cytoadhesins, cytokines, tissue factor expression) of ECs will be examined. Susceptibility of ECs to SARS-COV-2 infection will be determined.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients: age > 18 yr
* SARS-COV-2 infection within 12 months and positive lupus anticoagulant
* Patients with cardiovascular risk factors: at least among
* Hypertension, Dyslipidemia, Diabetes mellitus, obesity, smoker, Healthy volunteers

Exclusion Criteria:

* Significant comorbidities (active cancer, auto-immune diseases…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Covid-19 patients
  * patients with coronary artery disease
  * healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Western blot measurement of ACE2 receptor expression in porcine cells | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Olivier MOREL, Strasbourg, France